CLINICAL TRIAL: NCT01466686
Title: A Phase II Trial of Low Dose Fractionated Radiation Therapy as a Chemo-Potentiator of Salvage Temozolomide for Recurrent Anaplastic Astrocytoma and Glioblastoma Multiforme
Brief Title: Low Dose Radiation Therapy for Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J11120; NA_00065863 (Other: Johns Hopkins University School of Medicine)
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: High Grade Glioma
Keywords: Recurrent Glioblastoma Multiforme; Recurrent Anaplastic Astrocytoma; Surgery; Adjuvant Radiation; Adjuvant Temozolomide
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide with Low Dose Fractionated Radiation Therapy (Experimental): All patients will receive temozolomide (150 to 200 mg per square meter for 5 days during each 28 day cycle) for a total of 1 year or until the time of disease progression.
  All patients will receive 0.5 Gy of radiation therapy twice daily. This study will include a safety run-in component. If > 33% of patients in the initial cohort of 6 experience grade 3 or greater hematologic toxicity according to the NCI Common Toxicity Criteria version 4, then a dose reduction will occur following the schedule listed below. Otherwise, following a 1 month waiting period after the first cycle of adjuvant LDFRT plus temozolomide for the first cohort of patients, the phase 2 study will open for full accrual. Patients will receive radiation with the first six 28-day cycles of temozolomide.
  Interventions: Radiation: Low Dose Fractionated Radiation Therapy (LDFRT); Drug: Temozolomide

INTERVENTIONS:
Radiation: Low Dose Fractionated Radiation Therapy (LDFRT) — All patients will receive 0.5 Gy of radiation therapy twice daily. This study will include a safety run-in component. If > 33% of patients in the initial cohort of 6 experience grade 3 or greater hematologic toxicity according to the NCI Common Toxicity Criteria version 4, then a dose reduction will occur following the schedule listed below.
Drug: Temozolomide — All patients will receive temozolomide (150 to 200 mg per square meter for 5 days during each 28 day cycle) for a total of 1 year or until the time of disease progression.

SUMMARY:
To evaluate the safety and effectiveness of low dose rate radiation therapy plus temozolomide. This will be in patients with High Grade Glioma (to only include Anaplastic Astrocytoma or Glioblastoma Multiforme) who have previously been treated with surgery followed by radiation surgical resection followed by adjuvant radiation therapy plus temozolomide.

DETAILED DESCRIPTION:
In vitro and in vivo studies have suggested that low dose fractionated radiation therapy (LDFRT) may be used to potentiate full dose chemotherapy, decreasing the development of resistance found with standard doses of radiation and chemotherapy. This is a nonrandomized, open label, single institution phase II trial with a safety run-in to evaluate the safety and efficacy of LDFRT plus temozolomide in patients with High Grade Glioma (to only include Anaplastic Astrocytoma or Glioblastoma Multiforme) previously treated with surgical resection followed by adjuvant radiation therapy plus temozolomide. The primary objective of the phase II study is to estimate response rate in patients treated with twice daily fractions of low dose radiation plus temozolomide chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent GBM (Glioblastoma Multiforme)or Anaplastic Astrocytoma.
* The diagnosis of GBM or Anaplastic Astrocytoma.
* Patients must have been previously treated with surgical resection (any extent okay) and adjuvant radiation therapy plus temozolomide.
* Patients must be at least 12 months from completion of radiation therapy
* At least 2 months from completion of temozolomide (to be consistent with the the "rechallenge" group from Perry et al. JCO 2010).
* Age >18 years
* ECOG performance status <2 (Karnofsky >60%, see appendix A).
* There must be measurable disease on MRI.
* Patients must have normal organ and marrow function as defined below:
* Women must not be pregnant
* Ability to understand and the willingness to sign a written informed consent document
* Temozolomide re-treatment is planned by the treating neuro-oncologist.
* The most recent brain tumor pathology obtained for the patient must be glioblastoma.

Exclusion Criteria:

* Must be able to receive an MRI
* Patients may not be receiving any other investigational cancer treatment agents at the time of enrollment.
* Patients may not have previously failed treatment with salvage temozolomide.
* Patients may not have previously failed treatment with a VEGF inhibitor.
* Patients may not have previously been treated with >1 course of radiotherapy.
* Patients may not have previously been treated with radiosurgery to the brain.
* Uncontrolled intercurrent illness
* Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use and acceptable method of birth control to avoid pregnancy for the entire study period and up to 12 weeks after the study are excluded. Male subjects must also agree to use effective contraception for the same period as above.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Redmond, M.D., Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient enrolled in the study and then chose to withdraw prior to assignment/treatment. No data was collected for that participant.
Groups:
- Temozolomide With Low Dose Fractionated Radiation Therapy: All patients will receive temozolomide (150 to 200 mg per square meter for 5 days during each 28 day cycle) for a total of 1 year or until the time of disease progression.
  All patients will receive 0.5 Gy of radiation therapy twice daily. This study will include a safety run-in component. If > 33% of patients in the initial cohort of 6 experience grade 3 or greater hematologic toxicity according to the NCI Common Toxicity Criteria version 4, then a dose reduction will occur following the schedule listed below. Otherwise, following a 1 month waiting period after the first cycle of adjuvant LDFRT plus temozolomide for the first cohort of patients, the phase 2 study will open for full accrual. Patients will receive radiation with the first six 28-day cycles of temozolomide.
  Low Dose Fractionated Radiation Therapy (LDFRT): All patients will receive 0.5 Gy of radiation therapy twice daily. This study will include a safety run-in component. If > 33% of patients in the initial cohort of 6 experience grade 3 or greater hematologic toxicity according to the NCI Common Toxicity Criteria version 4, then a dose reduction will occur following the schedule listed below.
  Temozolomide: All patients will receive temozolomide (150 to 200 mg per square meter for 5 days during each 28 day cycle) for a total of 1 year or until the time of disease progression.
Period: Overall Study
Arm/Group | Temozolomide With Low Dose Fractionated Radiation Therapy
Started | 31
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide With Low Dose Fractionated Radiation Therapy
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 53.74 [38.77 to 70.39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 27
  black | 2
  other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
met baseline criteria per protocol [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: To estimate the response rate to salvage temozolomide plus LDFRT.
Time Frame: 3, 6 and 12 month follow-up after therapy has been completed
Population: This data was not collected
Arm/Group | Temozolomide With Low Dose Fractionated Radiation Therapy
Number analyzed (Participants) | 0

2. Primary Outcome: Overall Survival Rate
Description: Overall survival rate is calculated as the median number of months that patients were alive for the cohort
Time Frame: up to 12 months after completion of temozolomide (48 weeks of treatment)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide With Low Dose Fractionated Radiation Therapy
Number analyzed (Participants) | 30
months | 9.6 [7.0 to 15.4]

3. Secondary Outcome: Progression Free Survival Rate
Description: Progression free survival rate is calculated as the median number of months for the cohort until patient's disease worsened/progressed
Time Frame: up to 12 months after completion of temozolomide (48 weeks of treatment)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide With Low Dose Fractionated Radiation Therapy
Number analyzed (Participants) | 30
months | 7.3 [5.6 to 11.0]

4. Secondary Outcome: Number of Patients With Hematologic Toxicities
Description: The number of patients with grade 3+ hematologic toxicities.
Time Frame: Approximately every month from study start until 48 weeks, and then up to 12 months after completion of temozolomide at 3, 6, and 12 months follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide With Low Dose Fractionated Radiation Therapy
Number analyzed (Participants) | 30
Participants | 8

5. Secondary Outcome: Number of Patients With Neurologic Toxicity
Description: The number of patients with reported grade 3+ neurologic toxicities
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide With Low Dose Fractionated Radiation Therapy
Number analyzed (Participants) | 30
Participants | 6

ADVERSE EVENTS:
Time Frame: Approximately every month from study start until 48 weeks, and then up to 12 months after completion of temozolomide at 3, 6, and 12 months follow up
Description: Other (Not Including Serious) Adverse Events data was not collected.
Arm/Group | Temozolomide With Low Dose Fractionated Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 28/30
Serious Adverse Events (participants affected / at risk) | 30/30
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide With Low Dose Fractionated Radiation Therapy (N=30)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 — Grade NS
Death (Disease Progression) (General disorders) | 19 — Grade 5
Death (NOS) (General disorders) | 4 — Grade 5
Aphasia (Nervous system disorders) | 1 — Grade 4
Disease Progression (General disorders) | 6 — Grade 4
Fatigue (General disorders) | 1 — Grade 4
Intraparenchymal Hemorrhage of Brain (Nervous system disorders) | 1 — Grade 4
Lymphocyte Count Decrease (Investigations) | 1 — Grade 4
Personality/Behavioral CTC (Psychiatric disorders) | 1 — Grade 4
ALT increased (Investigations) | 2 — Grade 3
Ambulatory Dysfunction / Inability to Walk (Nervous system disorders) | 2 — Grade 3
Aphasia (Nervous system disorders) | 1 — Grade 3
Bowel Incontinence (Gastrointestinal disorders) | 1 — Grade 3
Cognitive Disturbance (Psychiatric disorders) | 3 — Grade 3
Disease Progression (General disorders) | 4 — Grade 3
DVT (NOS) (Vascular disorders) | 2 — Grade 3
DVT (RLE) (Vascular disorders) | 1 — Grade 3
Fatigue (General disorders) | 3 — Grade 3
Headache (Nervous system disorders) | 1 — Grade 3
Hyperglycemia / Elevated Glucose (Metabolism and nutrition disorders) | 2 — Grade 3
Leukocytosis (Blood and lymphatic system disorders) | 1 — Grade 3
Lymphocyte Count Decreased (Investigations) | 6 — Grade 3
Lymphopenia (Investigations) | 1 — Grade 3
Memory Loss (Nervous system disorders) | 1 — Grade 3
Motor Neuropathy (Nervous system disorders) | 2 — Grade 3
Nausea (Gastrointestinal disorders) | 1 — Grade 3
Ocular-Visual (Eye disorders) | 1 — Grade 3
Pain (knee) (Musculoskeletal and connective tissue disorders) | 1 — Grade 3
Pain (lower back) (Musculoskeletal and connective tissue disorders) | 1 — Grade 3
Pain (NOS) (General disorders) | 1 — Grade 3
Platelet Count Decreased (Investigations) | 1 — Grade 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 — Grade 3
Seizure (Nervous system disorders) | 2 — Grade 3
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 3
Speech Impairment (Nervous system disorders) | 2 — Grade 3
Status Epilepticus (Nervous system disorders) | 1 — Grade 3
Tinnitus (Ear and labyrinth disorders) | 1 — Grade 3
Urinary Incontinence (Renal and urinary disorders) | 1 — Grade 3
Weakness (lower extremity) (Musculoskeletal and connective tissue disorders) | 3 — Grade 3
Weakness (NOS) (Musculoskeletal and connective tissue disorders) | 1 — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT01466686/Prot_SAP_000.pdf